CLINICAL TRIAL: NCT07322575
Title: Evaluation of TMAO Production in Human Body From High-carnitine Diet by Fecal Gbu Gene Testing
Brief Title: Development of Microbial Metabolism Gene Tests for Facilitating Precision Health and Preventive Medicine-Evaluation of TMAO Production in Human Body From High-carnitine Diet by Fecal Gbu Gene Testing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202507141RINB
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Gut Dysbiosis for TMAO Production From Red Meat Consumption
Keywords: TMAO; red meat; carnitine; gut microbiota; gbu gene cluster; cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Red Meat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Red meat tolerance test (Experimental): Participants are required to take 900 grams of beef in a meal. Before the intervention, participants are asked to dietary record two day before the intervention. Fecal samples will be collected before and after the intervention. Blood sample will be collected in 0hr, 24hr, 48hr after the intervention. Each participant needs to complete a food frequency questionnaire.
  Interventions: Other: Beef

INTERVENTIONS:
Other: Beef — 900 grams of lean beef

SUMMARY:
The risk of cardiovascular diseases from red meat consumption varies among individuals due to variations in gut microbiota. L-carnitine in red meat can be converted to Trimethylamine n-oxide (TMAO) in the body by certain bacteria. Not everyone experiences a significant increase in TMAO levels after consuming carnitine. Gut microbiota differences are observed between high and low TMAO producers. The presence of the γ-butyrobetaine utilization (gbu) gene in gut microbiota is linked to TMAO production. This clinical research aims to determine if the gbu gene can predict TMAO levels after intaking a large amount of red meat.

DETAILED DESCRIPTION:
The risk of developing cardiovascular diseases due to the consumption of red meat varies among individuals, and this may be attributed to differences in the composition and function of gut microbiota. Studies have found that red meat, rich in L-carnitine, may be metabolized by certain anaerobic bacteria in the intestines to produce trimethylamine N-oxide (TMAO) in the human body. Previous research utilizing the oral carnitine challenge test (OCCT) revealed that not everyone experiences a significant increase in blood TMAO levels after consuming carnitine. Moreover, individuals with high TMAO production and low TMAO production showed distinct differences in their gut microbiota.

Furthermore, we have discovered a significant correlation between the abundance of the gbu gene in gut microbiota and the production of TMAO in response to dietary carnitine intake. Therefore, through the design of clinical research, we aim to investigate and assess whether the abundance of the gbu gene in gut microbiota can predict the levels of TMAO produced in the human body under a large amount of red meat consumption.

ELIGIBILITY:
Inclusion Criteria:

* Adult with age between 18 to 70
* Willing and capable of intaking a large amount of beef

Exclusion Criteria:

* Antibiotics use within one month
* L-carnitine supplement use within one month
* Chronic diarrhea
* Myasthenia gravis
* Parathyroid disorders
* Chronic kidney disease
* Epilepsy
* Severe anemia
* Severe cardiovascular diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Fecal gbu gene abundance measured by qPCR | up to 7-10 days
Blood TMAO level measured by LC-MS/MS | before intervention, 24hr, 48hr after intervention
Platelet aggregation of blood by Light Transmission Aggregometry | up to 7-10 days
Gut microbiome profiles measured by shotgun metagenome sequencing | up to 7-10 days

SECONDARY OUTCOMES:
Carnitine intake measured by 24hr dietary record | up to 7-10 days

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The data will be uploaded to be public when the research is published